CLINICAL TRIAL: NCT03133650
Title: A Phase I Trial of Vascular-Targeted Photodynamic Therapy in Esophagogastric Cancer Patients With Moderate to Severe Dysphagia
Brief Title: A Trial of a New Type of Photodynamic Therapy (VTP) in the Treatment of Patients With Cancer of the Esophagus Who Have Trouble Swallowing
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weizmann Institute of Science (Other); Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-319
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Esophagogastric Cancer; Moderate to Severe Dysphagia
Keywords: Vascular-Targeted Photodynamic Therapy (VTP); 15-319

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vascular-targeted photodynamic therapy (VTP) using WST11 (Experimental): Participants will receive intravenous administration of WST11 at a dose of 4 mg/kg, infused over 10 minutes, during an endoscopy procedure, followed by immediate laser light application.
  Interventions: Drug: WST 11-mediated VTP therapy

INTERVENTIONS:
Drug: WST 11-mediated VTP therapy — Administration of WST11 in conjunction with endoscopic illumination at 753 nm emitted by a diode laser and administered to the participant by optical fibre catheters (cylindrical light diffusers) and a standard upper GI endoscope.

SUMMARY:
The purpose of this study is to establish the highest dose of laser light for WST-11 VTP to treat obstruction from esophageal cancer that can be safely given.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Confirmed tissue diagnosis of esophageal squamous cell cancer, adenocarcinoma or poorly differentiated carcinoma, with pathology reviewed at MSKCC
* Has incurable disease defined as at least one of the following:

  * Presence of metastases to other organs (Stage IV), now or previously
  * Has locally advanced disease and are not candidates for surgery or more radiation treatment
  * Has received the maximal radiation therapy to the primary site, or has been assessed by radiation oncology as not being a candidate for chemoradiation therapy.
* Karnofsky performance status >/= 50%
* No endoluminal stent in place at the time of treatment
* Previous esophageal dilation is permitted, provided the patient has developed recurrent dysphagia since that procedure
* Patients should not have received any systemic therapy (including chemotherapy, biologic therapy or immunotherapy) </= 7 days prior to treatment
* Prior radiation or surgery to the esophagus is permitted for patients with locally recurrent/persistent disease
* Patients on prophylactic or full-dose anticoagulation are eligible, provided the treating physician believes it is safe to temporarily withhold anticoagulation (see Section 9.2)
* Adequate organ function defined at baseline as:

  * ANC ≥1,000/ L
  * Platelets ≥75,000/ L
  * Hb ≥8.5 g/dl
  * INR ≤1.5 (except for patients who are on full-dose warfarin)
  * Calculated creatinine clearance ≥50 ml/min (using Cockcroft-Gault method)
  * Total serum bilirubin ≤1.5 mg/dL, or </= 2.5 mg/dL for patients with a known history of Gilbert's syndrome
  * AST/ALT ≤5× upper limit of normal
* Able to provide written informed consent

Exclusion Criteria:

* Pregnant or breast-feeding women. Women of childbearing potential (WOCBP) must undergo a negative pregnancy test (either serum or urine) prior to study entry. Both sexes must use contraception while on study. WOCBP include:

  * Any woman who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation or oophorectomy) or who is not post-menopausal (defined as amenorrheic ≥12 consecutive months)
  * Women on hormone replacement therapy with documented serum follicle stimulating hormone level > 35 mIU/ml
  * Women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as intrauterine device or barrier methods to prevent pregnancy or are practicing abstinence of where the partner is sterile
* T4 tumors with involvement of any adjacent structure, including the trachea, aorta or pleura
* Prior history of esophageal perforation
* Any other medical or psychiatric comorbidities, including decompensated heart failure, unstable angina or coronary artery disease or severe pulmonary disease, that, in the opinion of the study investigator, would make the patient a poor candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated laser fluence rate | 60 days
  The maximally tolerated laser light fluence rate (mW/cm) of light exposure for VTP of malignant obstruction due to esophagogastric cancer will be measured by examining 6 fluence rates beginning with a fluence rate of 150 nW/cm, then increasing by 50mW/cm, up to a maximum of 400 mW/cm (150, 200, 250 300, 350, 400).

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gerdes, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (2):
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center (Data Analysis Only), New York, New York
- Weizmann Institute of Science, Rehovot, Israel

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/